CLINICAL TRIAL: NCT00297557
Title: Dual Time Point PET Imaging in Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: CCR2733
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-01

CONDITIONS: Hodgkin's or Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Comparison of single time point with dual time point PET imaging in the accuracy of diagnosing active lymphoma. Biopsy results or clinical/radiological progression will be used in conjunction with the PET data.

ELIGIBILITY:
Inclusion Criteria:

- Age 16 and above Diagnosis of Hodgkin's or Non-Hodgkin's lymphoma PET scan scheduled as part of management

Exclusion Criteria:

* Pregnant or lactating Diabetes mellitus

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gary Cook, Principal Investigator — Royal Marsden NHS Foundation Trust